CLINICAL TRIAL: NCT07268014
Title: The Effect of Pelvic Floor Exercises During Pregnancy on Obstetric Outcomes and Urinary Incontinence: A Prospective Randomized Controlled Trial
Brief Title: Effects of Pelvic Exercises on Birth and Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Assoc. Prof. Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/1051
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Maternal-Fetal Relations; Birth, First; Incontinence, Urinary; Pelvic Floor Disorders
Keywords: Pelvic Floor Exercise; Obstetric Outcomes; Urinary Incontinence; Birth, First
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (Placebo Comparator): The control group will consist of pregnant women who do not do any pelvic floor exercises.
  Interventions: Other: Pelvic Exercise Group
- Intervention Group (Experimental): Pregnant women in the exercise group will participate in an eight-week pelvic floor exercise program. The program begins with a face-to-face group training session during a childbirth preparation class at Konya City Hospital, in groups of 15, led by a midwife. Training covers pelvic floor anatomy, correct muscle identification, Kegel exercises, breathing, relaxation techniques, and exercise demonstrations.
  Following the session, participants will perform exercises three times a week for eight weeks, including Kegels, breathing-coordinated contractions, pelvic floor exercises in various positions, core stabilization exercises, and integration into daily activities. Weekly video materials will support proper exercise and motivation, and participants will record their practice in an exercise diary. At the end, experiences will be evaluated, and guidance for postpartum continuation will be provided.
  Interventions: Other: Pelvic Exercise Group

INTERVENTIONS:
Other: Pelvic Exercise Group — Pregnant women in the exercise group will participate in an eight-week pelvic floor exercise program. The program begins with a face-to-face group training session during a childbirth preparation class at Konya City Hospital, in groups of 15, led by a midwife. Training covers pelvic floor anatomy, correct muscle identification, Kegel exercises, breathing, relaxation techniques, and exercise demonstrations.
  Following the session, participants will perform exercises three times a week for eight weeks, including Kegels, breathing-coordinated contractions, pelvic floor exercises in various positions, core stabilization exercises, and integration into daily activities. Weekly video materials will support proper exercise and motivation, and participants will record their practice in an exercise diary. At the end, experiences will be evaluated, and guidance for postpartum continuation will be provided.

SUMMARY:
The Effect of Pelvic Floor Exercises During Pregnancy on Obstetric Outcomes and Urinary Incontinence: A Prospective Randomized Controlled Trial

DETAILED DESCRIPTION:
The study is a randomized controlled trial. It will be conducted at Konya City Hospital between December 2025 and June 2026. A total of 151 primiparous pregnant women will be included in the study (intervention group n=75, control group n=76). The intervention group will receive a pelvic floor exercise program, while the control group will not perform any pelvic floor exercises. Data will be collected using a personal information form, a pre-labor and post-labor follow-up form, and the Michigan Incontinence Severity Index.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the hospital's prenatal school and actively participating in the 3-day training sessions,
* Aged between 18 and 35 years,
* Between 28 and 30 weeks of gestation,
* Having a singleton and low-risk pregnancy,
* Primiparous (expecting their first birth),
* Voluntarily agreeing to participate by signing the written informed consent form,
* Able to read, understand, and communicate in Turkish.

Exclusion Criteria:

* Those who have previously given birth vaginally or by cesarean section (multiparous women),
* Those with multiple pregnancies,
* Those who conceived through assisted reproductive techniques,
* Those diagnosed with serious obstetric or medical complications during pregnancy (e.g., preeclampsia, gestational diabetes, risk of preterm birth),
* Those with chronic constipation or cough,
* Those who are overweight or obese,
* Those with chronic or recurrent urinary tract infections,
* Those with a history of psychiatric diagnosis or currently receiving psychiatric treatment,
* Those with a diagnosis of or treatment for urinary incontinence,
* Those unable to regularly attend the education sessions or who discontinue the program,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the sociodemographic characteristics of pregnant women before the training with a survey. | 7 month
  Sociodemographic information of pregnant women will be collected through surveys, compared, and reported.
Comparison of obstetric characteristics of pregnant women before the training with a questionnaire. | 7 month
  Obstetric data of pregnant women will be collected through questionnaires, compared, and reported.
Comparison of delivery methods among pregnant women across groups. | 7 month
  Labor and postpartum data will be collected, compared, and reported using a follow-up form.
Comparison of the severity of episiotomy in pregnant women between groups. | 7 month
  Pregnancy and postpartum follow-up data will be collected, compared, and reported using a form.
Comparison of the Michigan Incontinence Severity Index for pregnant women between groups. | 7 month
  The Michigan Incontinence Severity Index (M-ISI) will be administered to pregnant women. The scale consists of three subscales: stress incontinence, urge incontinence, and pad use/discomfort. Each subscale is scored separately. The RM-ISI ranges from 0 to 40 points (min-max), a higher score indicates more severe symptoms/discomfort for the relevant subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Seyhan Çankaya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No